CLINICAL TRIAL: NCT02183064
Title: A Multi-Center, Randomized, Parallel-Group, Open-Label Study to Compare Prescription Non-Steroidal Anti-Inflammatory Drug (NSAID) Changes, Health Care Utilization, Efficacy and Safety of Meloxicam 7.5 mg Versus Usual Care Administration of Prescription NSAIDs in a Managed Healthcare Setting in Patients With Osteoarthritis of the Hip, Knee, Hand or Spine
Brief Title: Study to Compare Prescription Non-Steroidal Anti-Inflammatory Drug (NSAID) Changes, Health Care Utilization, Efficacy and Safety of Meloxicam 7.5 mg Versus Usual Care Administration of Prescription NSAIDs in a Managed Healthcare Setting in Patients With Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107.210
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Meloxicam; Anti-Inflammatory Agents, Non-Steroidal

ARMS (2):
- Meloxicam (Experimental)
  Interventions: Drug: Meloxicam
- Usual care prescription NSAID (Active Comparator)
  Interventions: Drug: NSAID

INTERVENTIONS:
Drug: Meloxicam
  Arms: Meloxicam
Drug: NSAID
  Arms: Usual care prescription NSAID

SUMMARY:
Study to compare the percentage of treatment successes or failures in patients randomized to meloxicam 7.5 mg vs. usual care prescription NSAIDs. Additionally, health care utilization, efficacy and safety of patients in a managed healthcare setting with osteoarthritis (OA) of the hip, knee, hand or spine will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over the age of 18
* The patient, if female and of reproductive potential (i.e. neither surgically sterilized nor post-menopausal), must be practicing adequate contraception (e.g. intrauterine device, contraceptive pills, Depo-Provera, or implant or double barrier device) for at least three months prior to and for the duration of their trial participation and must have a negative pregnancy test at screening. Abstinence is not considered to be an acceptable method of contraception. (It should be noted that NSAIDs might interfere with the effectiveness of intrauterine devices)
* The patient must have a documented diagnosis of at least one of the following:

  * Osteoarthritis of the hip
  * Osteoarthritis of the knee
  * Osteoarthritis of the hand or
  * Osteoarthritis of the spine - Patients must have radiographic confirmation of the diagnosis
* The patient is willing to change or requires a change in current prescription NSAID therapy or requires initiation of prescription NSAID therapy for treatment of OA of the hip, knee, hand or spine
* The patient intends to remain a member of their present Managed Care Organization (MCO) for the duration of the trial
* The patient is willing to comply with instructions and to provide written informed consent

Exclusion Criteria:

* The patient has a known or suspected hypersensitivity to the trial drugs or their excipients, analgesics, antipyretics or NSAIDS (prescription or over-the-counter)
* The patient has received an investigational drug or used an investigational device within 30 days prior to entering the trial
* In the opinion of the investigator the patient has any disease or condition that may result in altered absorption, excess accumulation or impaired metabolism or excretion of the trial medication
* The patient has a history of recurrent peptic ulcer or history (within the past 6 months) of gastrointestinal perforation, peptic ulceration documented by endoscopy or radiography, symptomatic hiatal hernia requiring daily treatment or any history of a gastrointestinal tract hemorrhage, except simple hemorrhoidal bleeding
* The patient is currently on coumadin or might be placed on coumadin during the course of the clinical trial
* Patients with dementia, i.e. incapable of following directions or complying with the study protocol
* Patients with co-existing rheumatological disorders including rheumatoid arthritis
* The patient has previously participated in this trial
* Patients with coexisting fibromyalgia or ankylosing spondylitis
* Patient is pregnant or lactating
* Patient has severe hepatic failure
* Patient has non-dialysed renal failure
* Patient has history of GI bleed within the past 6 months
* Patient has history of cerebrovascular bleeding or other bleeding disorders
* Patient is receiving concomitant lithium, heparin or ticlopidine therapy
* Patient has a history of leukopenia (White Blood Cell count < 3500/mm³)
* The patient has a history of platelet count below the lower limit of normal or has a documented abnormal prothrombin time (PT) or partial thromboplastin time (PTT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1309 (Actual)
Dates: Start 1998-10; Primary Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Percentage of treatment successes and failures in patients randomized to meloxicam 7.5 mg vs.usual care prescription NSAIDs | up to 6 month

SECONDARY OUTCOMES:
Investigator's Global Assessment of Disease Activity (Likert) | Screening (Day 0), after six month (Day 180)
Patient's overall Assessment of pain over the past week on a visual analogue scale (VAS) | Day 0, 30, 60, 90, 120, 150, 180
Patient's Assessment of Health Status (VAS) | Day 0, 30, 60, 90, 120, 150, 180
Patient's Assessment of Satisfaction of Health | Day 0, 30, 60, 90, 120, 150, 180
Utility Index (VAS) | Day 0, 30, 60, 90, 120, 150, 180
Western Ontario and Mc Master University Osteoarthritis Index (WOMAC) | Day 0, 30, 60, 90, 120, 150, 180
Medication Compliance | Day 30, day 180
Disability Index | Screening (Day 0), after six month (Day 180)
Permanent Discontinuation of Study Medication related to lack of efficacy | up to day 180
Incidence and intensity of adverse events | from day 30 until day 180
Permanent Discontinuation of Study Medication related to adverse event | from day 30 until day 180